CLINICAL TRIAL: NCT00887575
Title: Phase I/II Trial of Neoadjuvant Sunitinib Administered With Weekly Paclitaxel/Carboplatin in Patients With Locally Advanced Triple-Negative Breast Cancer
Brief Title: Neoadjuvant Sunitinib With Paclitaxel/Carboplatin in Patients With Triple-Negative Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 122
Record Dates: First submitted 2009-04-22; First posted 2009-04-24 (Estimated); Results first posted 2014-12-17 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Triple-Negative; Paclitaxel; Carboplatin; Sunitinib; Sutent; Neoadjuvant
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Carboplatin; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose Level I (Experimental): Neoadjuvant - Paclitaxel IV (70 mg/m^2) days 1, 8 and 15 of each cycle, Carboplatin IV (AUC = 5) day 1 of every cycle and Sunitinib PO (25mg) daily.
  Maintenance - Sunitinib PO (25mg) daily
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Sunitinib
- Dose Level II (Experimental): Paclitaxel IV (80 mg/m^2) days 1, 8 and 15 of each cycle, Carboplatin IV (AUC = 5) day 1 of every cycle and Sunitinib PO (25mg) daily.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Sunitinib
- Dose Level III (Experimental): Paclitaxel IV (80 mg/m^2) days 1, 8 and 15 of each cycle, Carboplatin IV (AUC = 6) day 1 of every cycle and Sunitinib PO (25mg) daily.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Sunitinib

INTERVENTIONS:
Drug: Paclitaxel — IV infusion per institutional guidelines on Days 1, 8 and 15 of a 28 day cycle as follows depending on dose level (DL): DL1- 70 mg/m2, DL2- 80 mg/m2, DL3- 80mg/m2, DL4- 80mg/m2, DL-1- 70mg/m2, DL-2- 60mg/m2
  Other Names: Taxol; Systemic Therapy
Drug: Carboplatin — IV infusion per institutional guidelines Day 1 of a 28 day cycle as follows depending on dose level (DL): DL1- AUC=5, DL2- AUC=5, DL3- AUC=6, DL4- AUC=6, DL-1- AUC=4, DL-2- AUC=4
  Other Names: Paraplatin; Systemic Therapy
Drug: Sunitinib — By mouth (PO) once daily on days 1-21 of a 28 day cycle as follows depending on dose level (DL): DL1- 25mg, DL2-25mg, DL3- 25mg, DL4- 37.5mg, DL-1- 25mg, DL-2- 25mg. Maintenance therapy of 25mg daily
  Other Names: Sutent; Systemic Therapy

SUMMARY:
This trial will examine the combination of sunitinib plus paclitaxel and carboplatin as neoadjuvant treatment for locally advanced breast cancer.

DETAILED DESCRIPTION:
This open label, Phase I/II trial is designed to evaluate the combination of sunitinib plus paclitaxel and carboplatin as neoadjuvant treatment for locally advanced breast cancer. The Phase I portion of this study will determine the maximum tolerated dose (MTD) of paclitaxel, sunitinib and carboplatin that can be used together as neoadjuvant treatment in patients with locally advanced breast cancer. The MTD identified in the Phase I portion of the study will be used in the Phase II portion which will evaluate the efficacy, safety, and tolerability of neoadjuvant sunitinib/paclitaxel/carboplatin given for 6 cycles in patients with locally advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients, age ≥18 years
2. Histologically confirmed invasive ER-, PR-, and HER2-negative (triple-negative) adenocarcinoma of the breast
3. Triple-negative tumors are defined as:

   * For HER2-negative:
   * Fluorescence in situ hybridization (FISH)-negative (defined by ratio <2.2) OR
   * Immunohistochemical (IHC) 0, IHC 1+, OR
   * IHC 2+ or IHC 3+ and FISH-negative (defined by ratio <2.2)
   * For ER- and PR-negative: <10% tumor staining by immunohistochemistry (IHC)
4. Primary palpable disease confined to a breast and axilla on physical examination. For patients without clinically suspicious axillary adenopathy, the primary tumor must be larger than 2 cm in diameter by physical exam or imaging studies (clinical T2-T3, N0-N1, M0). For patients with clinically suspicious axillary adenopathy, the primary breast tumor can be any size (clinical T1-3, N1-2, M0). T1N0M0 lesions are excluded. Patients with metastatic disease are excluded.
5. Patients without clearly defined palpable breast mass or axillary lymph nodes but radiographically measurable tumor masses are eligible. Accepted procedures for measuring breast disease are mammography, MRI, and breast ultrasound. Patients with lesions measurable only by imaging will require repeat imaging after 3 cycles and prior to surgery
6. Eastern Cooperative Oncology Group performance status (ECOG PS) 0-2
7. Neuropathy grade <1 by the Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v 3.0)
8. Resolution of all acute effects of surgical procedures to grade ≤1.

   For patients who had, or will have sentinel lymph node and/or axillary dissection prior to initiation of study treatment, completion at least 4 weeks prior to starting study treatment and well-healed wound is required
9. Adequate hematologic function with:

   * Absolute neutrophil count (ANC) >1500/μL
   * Platelets ≥100,000/μL
   * Hemoglobin ≥10 g/dL
10. Adequate hepatic and renal function with:

    * Serum bilirubin ≤ the institutional upper limit of normal (ULN)
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x institutional ULN
    * Alkaline phosphatase ≤2.5 x institutional ULN
    * Serum creatinine ≤1.5 x ULN or calculated creatinine clearance ≥40 mL/min
11. Left ventricular ejection fraction (LVEF) ≥50% by multigated acquisition (MUGA) or echocardiogram (ECHO)
12. Bilateral, synchronous breast cancer is allowed if one primary tumor meets the inclusion criteria
13. Knowledge of the investigational nature of the study and ability to provide consent for study participation
14. Ability and willingness to comply with study visits, treatment, testing, and other study procedures

Exclusion Criteria:

1. Previous treatment for this breast cancer
2. Previous treatment with paclitaxel or carboplatin
3. Previous treatment with sunitinib or other angiogenic inhibitors (including, but not limited to bevacizumab, sorafenib, thalidomide)
4. Any of the following within the 12 months prior to starting study treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, cerebrovascular accident including transient ischemic attack, or pulmonary embolus
5. Uncontrolled hypertension (blood pressure >150/100 mmHg despite optimal medical therapy)
6. Ongoing cardiac dysrhythmias grade ≥2, atrial fibrillation of any grade, or prolongation of the QTc interval to >470 msec
7. Major surgery, significant traumatic injury, or radiation therapy within 4 weeks of starting study treatment. An interval of at least 1week is required following minor surgical procedures, with the exception of placement of a vascular access device
8. Grade 3 hemorrhage within 4 weeks of starting study treatment
9. Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication
10. Known human immunodeficiency virus (HIV) infection or other serious infection
11. Concomitant treatment with drugs having proarrhythmic potential including terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, indapamide, and flecainide
12. Concurrent use of the potent CYP3A4 inhibitors ketoconazole, itraconazole, clarithromycin, atazanavir, nefazodone, saquinavir, telithromycin, ritonavir, amprenavir, indinavir, nelfinavir, delavirdine and voriconazole and CYP3A4 inducers rifampin, rifabutin, rifapentine, phenobarbital, phenytoin, carbamazepine, St. John's Wort, and dexamethasone. Use of dexamethasone for study premedication is allowed. Grapefruit and grapefruit juice is prohibited. Alternative therapies should be used when available. If use of a potent CYP3A4 inhibitor or inducer is necessary, this must be approved by the Study Chair
13. Known or suspected hypersensitivity to drugs containing Cremophor®EL (polyoxyethylated castor oil) such as cyclosporine or teniposide
14. Pregnancy or breast-feeding. Negative serum pregnancy test is required within 7 days prior to first study treatment (Day 1, Cycle ) for all women of childbearing potential. Patients of childbearing potential must agree to use a birth control method that is approved by their study physician while receiving study treatment and for three months after the last dose of study treatment. Patients must agree to not breast-feed while receiving study treatment
15. Concurrent treatment with an ovarian hormonal replacement therapy or with hormonal agents such as raloxifene, tamoxifen or other selective estrogen receptor modulator (SERM). Patients must have discontinued use of such agents prior to beginning study treatment
16. History of malignancy treated with curative intent within the previous 5 years with the exception of skin cancer, cervical carcinoma in situ, or follicular thyroid cancer. Patients with previous invasive cancers (including breast cancer) are eligible if the treatment was completed more than 5 years prior to initiating current study treatment, and there is no evidence of recurrent disease
17. Use of any investigational agent within 30 days of administration of the first dose of study drug or concurrent treatment on another clinical study
18. Requirement for radiation therapy concurrent with study anticancer treatment. Patients who require breast or chest wall radiation therapy after surgery are eligible, but will have maintenance sunitinib interrupted while receiving radiation
19. Any other disease(s), psychiatric condition, metabolic dysfunction, or findings from a physical examination or clinical laboratory test result that would cause reasonable suspicion of a disease or condition, that contraindicates the use of study drugs, that may increase the risk associated with study participation, that may affect the interpretation of the results, or that would make the patient inappropriate for this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-06; Primary Completion 2013-07 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise A Yardley, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (14):
- United States (14):
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Florida Cancer Specialists North, Fort Myers, Florida
  - Florida Cancer Specialists South, Fort Myers, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Providence Medical Group, Terre Haute, Indiana
  - Baptist Hospital East, Louisville, Kentucky
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - National Capital Clinical Research Consortium, Bethesda, Maryland
  - St. Louis Cancer Care, Chesterfield, Missouri
  - Nebraska Methodist Cancer Center, Omaha, Nebraska
  - Hematology Oncology Associates of Northern NJ, Morristown, New Jersey
  - Cancer Centers of Southwest Oklahoma, Lawton, Oklahoma
  - Family Cancer Center, Collierville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at multiple dose levels into the Dose Escalation (Phase I) portion of this study to determine the safest dose of this regimen (MTD- Maximum Tolerated Dose). Upon determination of this dose, patients being treated at the MTD proceeded to the Dose Expansion (Phase II) portion of the study and additional patients were recruited
Period: Phase I
Arm/Group | Dose Level I | Dose Level II | Dose Level III
Started | 6 | 6 | 3
Completed | 6 | 0 (Patients were on-study until determination of the Maximum Tolerated Dose (MTD)) | 0 (Patients were on-study until determination of the Maximum Tolerated Dose (MTD))
Not Completed | 0 | 6 | 3
Period: Phase II - Neoadjuvant Therapy
Arm/Group | Dose Level I | Dose Level II | Dose Level III
Started | 41 (Includes patients treated at MTD during Phase I, 39 additional patients enrolled, 4 were not treated) | 0 | 0
Completed | 16 | 0 | 0
Not Completed | 25 | 0 | 0
Period: Phase II - Maintenance Therapy
Arm/Group | Dose Level I | Dose Level II | Dose Level III
Started | 8 (Pts who completed 6 cycles of Neoadjuvant Therapy & underwent surgery were eligible for maintenance) | 0 | 0
Completed | 6 | 0 | 0
Not Completed | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Between June 2009 and July 2012, 54 patients were enrolled (15 in phase I and 39 additional patients in phase II). Three patients were later found to be ineligible and were excluded from the analysis. An additional patient did not receive any study treatment and is also excluded from the analysis.
Groups:
- All Patients: Includes all patients treated at all dose levels
Arm/Group | All Patients
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: Years] | 53 [32 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 36
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 50
Baseline ECOG Performance Status [Number; unit: participants] — ECOG Performance Status = 0 - Asymptomatic (Fully active, able to carry on all predisease activities without restriction)
  ECOG Performance Status = 1 - Symptomatic but completely ambulatory (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. For example, light housework, office work)
  participants
    ECOG Performance Status = 0 | 45
    ECOG Performance Status = 1 | 5
Menopausal Status [Number; unit: Participants]
  Postmenopausal | 34
  Premenopausal | 16

OUTCOME MEASURES:

1. Primary Outcome: Phase II: The Number of Subjects Exhibiting Pathologic Complete Response to Neoadjuvant Treatment With Sunitinib/Paclitaxel/Carboplatin
Description: Pathologic complete response (PCR) is defined as no residual invasive breast cancer in final breast or axillary lymph node samples.
Time Frame: at weeks 26-30
Population: Patients treated at Dose Level I (Phase I and Phase II) who underwent surgery
Measure: Number; unit: participants
Groups:
- Phase II- Sunitinib/Paclitaxel/Carboplatin: Systemic Therapy based on maximum tolerated dose (MTD) of the Phase I portion
Arm/Group | Phase II- Sunitinib/Paclitaxel/Carboplatin
Number analyzed (Participants) | 32
participants | 12

2. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Assessments will be made through analysis of reported incidence of treatment-emergent adverse events (AEs) and serious adverse events (SAEs) at the phase II dose
Time Frame: Days 1, 8, and 15 of each 4-week cycle up to 24 weeks during neoadjuvant treatment, and every 4 weeks during maintenance treatment
Population: The safety analysis includes all eligible patients enrolled at the MTD, whether or not treatment was recieved (6 patients in Phase I were treated at the MTD, 39 patients were enrolled in Phase II, 3 were deemed ineligible after enrollment-thus 42 patients are included in the safety analysis, including 1 eligible patient who was not treated)
Measure: Number; unit: participants
Arm/Group | Phase II- Sunitinib/Paclitaxel/Carboplatin
Number analyzed (Participants) | 42
participants
  Neutropenia | 34
  Anemia | 30
  Thrombocytopenia | 30
  Leukopenia | 30
  Febrile neutropenia | 3
  Fatigue | 32
  Alopecia | 26
  Nausea/Vomiting | 24
  Constipation | 22
  Diarrhea | 21
  Mucositis | 17
  Dysgeusia | 17
  Peripheral neuropathy | 17
  Dyspepsia | 13
  Dyspnea | 12
  Anorexia | 10
  Fever | 9
  Bleeding | 9
  Insomnia | 9
  Pain in extremity | 9
  Skin toxicity | 9

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Assessed by clinical, radiologic and surgical determinations before and after neoadjuvant therapy. Measurable lesions will be defined by RECIST criteria v1.1.
Time Frame: Days 1, 8 and 15 of each cycle, minimum of 12 weeks
Population: Patients who were enrolled, treated at the MTD and completed at least 3 cycles of neoadjuvant therapy
Measure: Number; unit: participants
Arm/Group | Phase II- Sunitinib/Paclitaxel/Carboplatin
Number analyzed (Participants) | 29
participants | 25

4. Secondary Outcome: Disease-free Survival
Description: Defined as the time between day of surgery to first documented disease occurrence or death due to any cause.
Time Frame: every 4 weeks from date of surgery until treatment discontinuation or death, expected average 18 months
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Dose Level I
Number analyzed (Participants) | 41
months
  Median Overall Survival | NA [40.9692 to NA] — Not enough data available for this outcome measure
  Median Disease-Free Survival | 15.8357 [6.8665 to NA] — Not enough data available for this outcome measure

5. Secondary Outcome: Overall Survival (OS)
Description: Defined as the time between Day 1 Cycle 1 to time of death from any cause.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: probability of overall survival at 24 m
Arm/Group | Dose Level I
Number analyzed (Participants) | 41
probability of overall survival at 24 m | 0.8912 [0.7340 to 0.9580]

ADVERSE EVENTS:
Arm/Group | Dose Level I
Serious Adverse Events (participants affected / at risk) | 3/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level I (N=41)
ACUTE RENAL FAILURE (Renal and urinary disorders) | 1 (1)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
CREATININE LEVELS INCREASED (Investigations) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 1 (2)
DIZZINESS (Nervous system disorders) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1)
EDEMA (General disorders) | 1 (3)
FATIGUE (General disorders) | 2 (4)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 1 (1)
FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
HYPERMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (3)
MUCOSITIS (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (5)
PHARYNGITIS (Infections and infestations) | 1 (1)
TASTE ALTERATION (Nervous system disorders) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (3)
VOMITING (Gastrointestinal disorders) | 2 (3)
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level I (N=41)
ALANINE AMINOTRANSFERA (Investigations) | 3 (5)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 3 (5)
ALLERGIC REACTION (Immune system disorders) | 4 (8)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 4 (6)
ALOPECIA (Skin and subcutaneous tissue disorders) | 24 (79)
ANEMIA (Blood and lymphatic system disorders) | 34 (135)
ANOREXIA (Metabolism and nutrition disorders) | 11 (25)
ANXIETY (Psychiatric disorders) | 4 (17)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 8 (23)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 (7)
ASTHENIA (Musculoskeletal and connective tissue disorders) | 3 (9)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 (11)
BLURRED VISION (Eye disorders) | 4 (16)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 4 (6)
BREAST PAIN (Reproductive system and breast disorders) | 5 (12)
CHEST PAIN (General disorders) | 4 (8)
CONSTIPATION (Gastrointestinal disorders) | 20 (60)
COUGH (Respiratory, thoracic and mediastinal disorders) | 9 (23)
DEHYDRATION (Metabolism and nutrition disorders) | 4 (5)
DEPRESSION (Psychiatric disorders) | 3 (5)
DIARRHEA (Gastrointestinal disorders) | 20 (54)
DIZZINESS (Nervous system disorders) | 14 (30)
DRY MOUTH (Gastrointestinal disorders) | 4 (14)
DRY SKIN (Skin and subcutaneous tissue disorders) | 4 (6)
DYSGEUSIA (Nervous system disorders) | 6 (11)
DYSPEPSIA (Gastrointestinal disorders) | 10 (29)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 13 (33)
EDEMA (General disorders) | 3 (11)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 10 (25)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 4 (5)
FATIGUE (General disorders) | 34 (125)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 3 (4)
FEVER (General disorders) | 8 (12)
FLUSHING (Vascular disorders) | 5 (12)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3 (12)
GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 4 (5)
HEADACHE (Nervous system disorders) | 13 (28)
HOT FLASHES (Vascular disorders) | 3 (6)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 4 (12)
HYPERTENSION (Vascular disorders) | 7 (18)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 3 (4)
HYPOKALEMIA (Metabolism and nutrition disorders) | 4 (4)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 3 (4)
INSOMNIA (Psychiatric disorders) | 14 (42)
LEUKOPENIA (Blood and lymphatic system disorders) | 31 (106)
MEMORY IMPAIRMENT (Nervous system disorders) | 3 (6)
MUCOSITIS (Gastrointestinal disorders) | 16 (29)
MYALGIA (Musculoskeletal and connective tissue disorders) | 10 (31)
NAIL DISCOLORATION (Skin and subcutaneous tissue disorders) | 3 (4)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 5 (8)
NASAL DRAINAGE (Respiratory, thoracic and mediastinal disorders) | 5 (7)
NAUSEA (Gastrointestinal disorders) | 32 (93)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3)
NEUTROPENIA (Blood and lymphatic system disorders) | 38 (132)
ORAL PAIN (Gastrointestinal disorders) | 7 (9)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 (22)
PERIPHERAL NEUROPATHY (Nervous system disorders) | 18 (56)
PRURITUS (Skin and subcutaneous tissue disorders) | 6 (10)
Pain (General disorders) | 9 (10)
RASH (Skin and subcutaneous tissue disorders) | 11 (28)
SCALP PAIN (Skin and subcutaneous tissue disorders) | 3 (11)
SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 4 (6)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 3 (5)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 5 (6)
TASTE ALTERATION (Nervous system disorders) | 16 (55)
THROAT PAIN (Gastrointestinal disorders) | 3 (4)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 32 (107)
THROMBOEMBOLIC EVENT (Vascular disorders) | 3 (3)
VOMITING (Gastrointestinal disorders) | 8 (18)
WEIGHT LOSS (Investigations) | 3 (6)
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 4 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites